CLINICAL TRIAL: NCT06795815
Title: The Implementation of the Go Wish Game to Promote Advance Care Planning in Onco-hematologic Disease (Onco-hema Go Wish-ACP): Intervention Set up and Multicentre Feasibility Trial
Brief Title: The Implementation of the Go Wish Game to Promote Advance Care Planning in Onco- Hematologic Disease
Acronym: OHGW-ACP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OHGW-ACP
Record Dates: First submitted 2025-01-08; First posted 2025-01-28 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-01

CONDITIONS: Leukemia; Multiple Mieloma; Advanced Solid Tumors; Lymphoma; Oncology; Hematologic Diseases
Keywords: Advance Care Planning; Go Wish Game; Medical Oncology; Hematology; Oncology; Palliative Care; Experimental Design Study; Mixed Methods
MeSH Terms: conditions — Leukemia; Lymphoma; Neoplasms; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients affected by refractory lymphomas, or leukemia or myeloma multiple or advanced solid tumors (Experimental)
  Interventions: Other: Go Wish Game

INTERVENTIONS:
Other: Go Wish Game — The Go Wish Game (GWG) provides a simple tool, composed by 35 cards to identify individual priorities. GWG is welcomed as a first step in clarifying values and personal thoughts linked to the end of life. The GWG discussion will be divided into two meetings. During the first one, the physician instructs the patients and their caregivers on how the GWG works. The patient will be invited to divide the cards into three sets, labeling the content of the cards within each set as: Very important;more or less important and not important.
  This will be the base for the second meeting. During the second meeting - scheduled within one week - each category of card sets will be discussed with patients and their caregivers. The identification of the most relevant wishes or priorities of each patient will be incorporated into the individual therapeutic plan and the patient will be offered the option to make a formal ACP in the following 4 weeks.

SUMMARY:
This is a mixed-method, device-free and drug-free multicenter interventional study. The study aims at facilitating end-of-life conversations within the doctor-patient relationship through the use of the Go Wish Game (GWG) and supporting patients, their caregivers and healthcare professionals to complete Advance Care Panning documentation.

The GWG helps people clarify and identify their priorities, should they be affected by a chronic, disabling and potentially non-healing illness. In fact, the GWG consists of a small deck of cards, and on each card is a concrete action or situation that may be important to a person at the end of life.

The "Onco-hema Go wish-ACP" project aims to evaluate the feasibility of a Go Wish Game-based intervention with patients with refractory lymphoma, leukemia or multiple myeloma or advanced solid tumors with prognosis > 3 months.

In terms of secondary objectives, the study aims to.

* Evaluate and compare the intervention with hematology and oncology patients in terms of: - Other feasibility indicators; Involvement in CCP pathways; Quality of communication; Meaning of life; Impact on hope; through a series of questionnaires administered to patients and caregivers involved in the intervention
* Qualitatively assess the acceptability of the intervention in terms of recruitment and delivery with patients and caregivers through semi-structured interviews and with professionals through Focus Groups (FGs).
* To analyze the clinical records of enrolled patients in terms of: values and preferences; awareness of prognosis; end-of-life choices and shared decision-making on treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years age; diagnosed with refractory lymphomas, or leukemia or multiple myeloma or advanced solid tumors and estimated prognosis > 3 months;
* able to communicate in Italian and
* to give written consent to the study.

Exclusion Criteria:

* Patients with severe cognitive impairment or serious psychiatric condition;
* refusal to participate to the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility | 1 Year
  We will evaluate the feasibility of the intervention. Feasibility will be investigated by:
  1. proportion of patients who will accept to participate among those screened/eligible who received the proposal to participate;
  2. proportion of enrolled patients who will withdraw from the study after the first GWG discussion among the enrolled patients; 3, percentage proportion of enrolled patients who will attend all the planned GWG discussions;
  4. proportion of enrolled patients that will complete the ACP document (after participating in all the planned GWG discussions)

SECONDARY OUTCOMES:
ACP Engagement; | 18 Months
  We will further assess and compare the intervention within hemato-oncological and oncological patients in terms of:
  1. ACP engagement: we will use the 4-item ACP Engagement (4-item ACP-E) questionnaire
Quality of Communication; | 18 Months
  We will further assess and compare the intervention within hemato-oncological and oncological patients in terms of:
  2. Quality of communication: we will use the 19-item Quality of Communication (QOC) questionnaire
Meaning of Life; | 18 Months
  We will further assess and compare the intervention within hemato-oncological and oncological patients in terms of:
  3. Meaning of life: we will use the Meaning in Life scale (MLS)
Impact on patients' hope | 18 Months
  We will further assess and compare the intervention within hemato-oncological and oncological patients in terms of:
  4. Impact on patients' hope: we will use the Hope Herth Index (HHI)
Acceptability | 18 Months
  5. Acceptability of intervention in terms of recruitment and intervention delivery will be further investigated by: semi-structured interviews with patients and caregivers and FG with HPs who applied the GWG.
  .
ACP documentation | 18 Months
  We will analyze the ACP documentation of patients enrolled to qualitatively investigate the congruence and relations between the priorities defined during the GWG meetings and the decisions written in the care plan

CONTACTS AND LOCATIONS:
Locations (1):
- AziendaUSL IRCCS Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: Yes
We share individual information about gender, age, work occupation, disease type, prognosis and time of diagnosis.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Access Criteria: The access will be able only to those people in terms of clinical staff, who are involved in the study